CLINICAL TRIAL: NCT00192465
Title: A Phase I, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI-524 (NUMAX TM), a Humanized Enhanced Potency Monoclonal Antibody Against Respiratory Syncytial Virus (RSV), in Healthy Adults
Brief Title: Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI-524 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Genevieve Lonosky, M.D., MedImmune Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MI-CP101
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — motavizumab

ARMS (5):
- 1 (Experimental): MEDI-524 (Numax-TM)
  Interventions: Biological: MEDI-524 (Numax-TM)
- 2 (Experimental): MEDI-524 (Numax-TM)
  Interventions: Biological: MEDI-524 (Numax-TM)
- 3 (Experimental): MEDI-524 (Numax-TM)
  Interventions: Biological: MEDI-524 (Numax-TM)
- 4 (Experimental): MEDI-524 (Numax-TM)
  Interventions: Biological: MEDI-524 (Numax-TM)
- 5 (Experimental): MEDI-524 (Numax-TM)
  Interventions: Biological: MEDI-524 (Numax-TM)

INTERVENTIONS:
Biological: MEDI-524 (Numax-TM) — Grp.1: 3 mg/kg IV (single dose)
  Arms: 1
Biological: MEDI-524 (Numax-TM) — Grp. 2: 15 mg/kg IV (single dose)
  Arms: 2
Biological: MEDI-524 (Numax-TM) — Grp. 3: 30 mg/kg IV (single dose)
  Arms: 3
Biological: MEDI-524 (Numax-TM) — Grp. 4: 3 mg/kg IM (single dose)
  Arms: 4
Biological: MEDI-524 (Numax-TM) — Grp.5: 3 mg/kg IM (two doses)
  Arms: 5

SUMMARY:
To provide safety, tolerability, pharmacokinetic, and immunogenicity data for MEDI-524 administered initially as a single dose to healthy adults in a dose escalation safety study before testing in the targeted pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must meet all of the following criteria:
* Age 18 through 49 years at the time of administration of study drug
* Weight £90 kg
* Healthy by medical history and physical examination
* Normal electrocardiogram (EKG) at screening (must be within 21 days before entry into the study)
* Written informed consent obtained from the volunteer
* Sexually active females, unless surgically sterile, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 14 days prior to the administration of study drug, must agree to continue using such precautions for 30 days after administration of study drug, and must have a negative serum pregnancy test within 7 days prior to the administration of study drug and a negative urine pregnancy test on the day of study drug administration.
* Ability to complete the follow-up period of 90 days (single-dose groups) or 120 days (two-dose group) as required by the protocol

Exclusion Criteria:

* Volunteers must have none of the following:
* Acute illness at the time of entry into the study
* Temperature ³99.5°F at the time of entry into the study
* Any drug therapy within 7 days prior to Study Day 0 (except for certain medications such as contraceptives, topical corticosteroids, or infrequent use of over-the-counter headache medications, following approval of the sponsor)
* Blood donation in excess of 400 mL within 6 months of the time of entry into the study
* Receipt of immunoglobulin or blood products within 60 days before entry into the study
* Receipt of any investigational drug therapy or standard vaccine within 120 days before administration of study drug in this protocol through 60 days after the final dose of study drug
* History of immunodeficiency or receipt of immunosuppressive drugs
* History of allergic disease or reactions likely to be exacerbated by any component of the study drug
* Previous medical history or evidence of an intercurrent illness that may compromise the safety of the volunteer in the study
* Evidence of any systemic disease on physical examination
* Evidence of infection with hepatitis A, B, or C virus or HIV-1
* At screening (must be within 7 days before study dose administration) any of the following: CBC: Hgb < 12.0 gm/dL; WBC < 4,000/mm3; platelet count < 120,000/mm3 (or laboratory normal values); AST, ALT, BUN, creatinine > upper limit of normal; other abnormal laboratory values in the screening panel which in the opinion of the principal investigator are judged to be clinically significant.
* Nursing mother
* History of alcohol or drug abuse within the past 2 years
* The presence of any condition or concern which in the opinion of the principal investigator may interfere with the conduct or interpretation of the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-11; Primary Completion 2004-04 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Safety | 30 days after patient's final dose of study drug
Pharmacokinetics | Study Day 0 and 60, 90 days after dose 1; and 7, 30, 60, 90 days after dose 2.
Immunogenicity | 150 days after final dose

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Losonsky, MD, Study Director — MedImmune LLC
Locations (1):
- SFBC International, Inc, Miami, Florida, United States